CLINICAL TRIAL: NCT01487369
Title: Special Survey of Production of Insulin Aspart (IAsp) Specific Antibody
Brief Title: Special Survey of Production of Insulin Aspart Specific Antibody
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1946
Record Dates: First submitted 2011-11-29; First posted 2011-12-07 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin Aspart
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Injected subcutaneously (s.c., under the skin). Prescribed by physician as a result of normal clinical practice.

SUMMARY:
This study is conducted in Japan. The aim of this study is to collect data of production of insulin aspart specific antibody under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes requiring insulin therapy

Exclusion Criteria:

* Patients who had a treatment history of NovoRapid® (insulin aspart)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes requiring insulin therapy and who had a treatment history of NovoRapid® (insulin aspart)
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2002-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Antibody titre findings

SECONDARY OUTCOMES:
Hypoglycemic events
Adverse events
HbA1c (glycosylated haemoglobin)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com